CLINICAL TRIAL: NCT00468793
Title: Randomized Clinical Study of Traditional Versus ScvO2 Guided Perioperative Fluid Therapy
Brief Title: Traditional Versus ScvO2 Guided Perioperative Fluid Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Gro Østgaard, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16312
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-05

CONDITIONS: Perioperative Care
Keywords: central venous saturation; bowel surgery; morbidity; intravenous infusions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Fluid therapy guided by blood pressure and urine production
  Interventions: Procedure: Intravenous fluid
- 1 (Experimental): ScvO2 guided fluid therapy
  Interventions: Procedure: Intravenous fluid

INTERVENTIONS:
Procedure: Intravenous fluid — The same intravenous fluids will be used in both arms but the volume will be different

SUMMARY:
Perioperative goal directed fluid therapy by means of an esophageal doppler has been shown to reduce morbidity and length of stay. In this study patients undergoing elective bowel surgery will be randomised to traditional fluid therapy with crystalloids versus fluid boluses guided by central venous oxygen saturation. The primary outcome will be complications after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective bowel surgery,
* Able to give informed consent

Exclusion Criteria:

* Coagulation defect,
* Renal failure,
* Valvular stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity | postoperative day 30

SECONDARY OUTCOMES:
serum creatinine | postoperative day 3

CONTACTS AND LOCATIONS:
Overall Officials: Gro Østgaard, M.D., PH.D., Study Chair — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway